CLINICAL TRIAL: NCT02040649
Title: Substudy of the NONSEDA-trial (NCT01967680): Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Me-chanical Ventilation - Effects on Posttraumatic Stress Disorder
Brief Title: Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Mechanical Ventilation - Effects on PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palle Toft (Other)
Collaborators: Kolding Sygehus (Other); The Danish Council for Strategic Research (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Palle Toft, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20130025b
Record Dates: First submitted 2014-01-10; First posted 2014-01-20 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Anxiety
Keywords: Critical care; Respiration, artificial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Respiratory Aspiration | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-sedation (Experimental): Non-sedation supplemented with pain management during mechanical ventilation.
  Interventions: Other: Non-sedation
- Sedation (Active Comparator): Current gold standard: Sedation with a daily wake-up trial.
  Interventions: Other: Control, sedation (propofol, midazolam)

INTERVENTIONS:
Other: Non-sedation — Patients are awake or have natural sleep during mechanical ventilation. Pain is treated with morphine iv.
  Arms: Non-sedation
Other: Control, sedation (propofol, midazolam) — Continuous iv-sedation (propofol first 48 hours, from then midazolam) to Ramsey 3-4 with a daily wake up attempt, where sedation is stopped until patient is awake.
  Arms: Sedation

SUMMARY:
Through many years, the standard care has been to use continuous sedation of critically ill patients during mechanical ventilation. However, preliminary randomised clinical trials indicate that it is beneficial to reduce the sedation level in these patients. The NONSEDA trial is an investigator-initiated, randomised, clinical, parallel-group, multinational, superiority trial designed to include 700 patients from at least six ICUs in Denmark, Norway and Sweden, comparing no sedation with sedation and a daily wake-up trial during mechanical ventilation. This is a substudy of the NONSEDA trial, concerning 250 patients included at trialsite Kolding, Denmark. The aim of the substudy is to assess the effects of no sedation on posttraumatic stress disorder after discharge from ICU.

Our hypothesis is that critically ill patients who are not sedated during mechanical ventilation will have less posttraumatic stress disorder after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheally intubated
* Expected time on ventilator > 24 hours
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Severe head trauma where therapeutic coma is indicated
* Therapeutic hypothermia where therapeutic coma is indicated
* Status epilepticus where therapeutic coma is indicated
* Patient has participated in the study before
* Patient is transferred from another ICU with length of stay > 48 hours
* Patient is comatose at admission
* PaO2/FiO2 ≤ 9, if sedation is necessary for oxygenation
* Patient does not speak Danish, swedish or norwegian at a reasonable level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
PTSD | 3 months after discharge from ICU
  Number of patients in each group diagnosed with PTSD by a neuropsycologist, based on an interview including posttraumatic stress disorder index and a general evaluation of the patient based on the ICD-10 criteria.

SECONDARY OUTCOMES:
Patient-reported quality of life | 3 months after discharge from ICU
  SF-36v2, mental component score for each group. The questionnaire is mailed to the participants, who complete it at home.
Depression | 3 months after discharge from ICU
  Number of patients in each group diagnosed with depresion by the neuropsycologist, based on personal interview and Beck depression inventory score.
Anxiety | 3 months after discarge from ICU
  Number of patients in each group diagnosed with anxiety by the neuropsycologist, based on personal interveiw and Beck anxiety inventory score.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Nedergaard, MD, Principal Investigator — Lillebaelt Hospital, Kolding
Locations (1):
- Lillebaelt Hospital, Kolding, Intensive Care Unit, Kolding, Denmark

REFERENCES:
- [Background] Strom T, Stylsvig M, Toft P. Long-term psychological effects of a no-sedation protocol in critically ill patients. Crit Care. 2011;15(6):R293. doi: 10.1186/cc10586. Epub 2011 Dec 13. PMID 22166673